CLINICAL TRIAL: NCT03904524
Title: SET-to-Meet; Pilot Testing of a Nurse-led Intervention to Ensure Routine Interdisciplinary Family Meetings in ICUs
Brief Title: SET-to-Meet; Pilot Testing of a Nurse-led Intervention
Acronym: SET-to-Meet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Cambia Health Foundation (Other)
Responsible Party: Principal Investigator, Jennifer Seaman, Assistant Professor, School of Nursing, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY18090002
Record Dates: First submitted 2019-03-27; First posted 2019-04-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Critical Illness
Keywords: Intensive Care Unit; Serious Illness Communication; Clinician-Family Communication; Family Support
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SET-to-MEET (Experimental): This is a single arm, open trial that will be conducted in parallel in 3 separate ICUs. Each site will receive the SET-to-MEET intervention.
  Interventions: Behavioral: SET-to-Meet

INTERVENTIONS:
Behavioral: SET-to-Meet — The overall objective of this study is to pilot test, in advance of a larger randomized trial, a scalable, nurse-led intervention to ensure timely interdisciplinary family meetings are held on behalf of critically-ill ICU patients who cannot participate in discussions about their care.

SUMMARY:
While interdisciplinary family meetings are evidence-based and part of usual care, this study seeks to test a novel set of implementation strategies (the SET-to-Meet intervention) to improve adherence to best practice guidelines for interdisciplinary family meetings. SET stands for Screen-Engage-Track; SET-to Meet is a nurse-led, team based intervention to ensure routine interdisciplinary family meetings are held on behalf of incapacitated, critically-ill patients in ICUs. This study is a feasibility and acceptability pilot test of the intervention.

DETAILED DESCRIPTION:
The intervention components are: a protocol for interdisciplinary family meetings that is tailored to the individual ICU unit and steps in the SET-to-Meet process: 1.) Screening of patients on admission to determine if patient meets criteria for a family meeting; 2.) proactively Engaging family members to inform them about the unit's protocol for family meetings and to find out who from the family might attend the meeting; and Tracking the progress of setting up the meeting (identifying the patient during ICU team rounds as a patient meeting criteria for a family meeting; discussing setting up the meeting with the ICU team; scheduling the meeting and communicating details to attendees.)

Implementation of the intervention includes: 1.) Working with the site ICU physician and nursing leadership to tailor the SET-to-meet protocol and tracking tool for family meetings, ensuring they are customized for the unit workflow and staffing model, and 2.) Providing on-line training and 2 weeks of on-site coaching to ICU nursing staff, care management/social work staff, and intensivists (MD and APP) in the use of the tailored protocol and tracking tool.

Feasibility and acceptability will be assessed by percentage of staff completing training, adherence to elements of the intervention, and number of patients meeting enrollment criteria. Acceptability will be assessed via focus groups and a survey testing satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Individuals ≥18 year of age, admitted to the ICU for intensive care services at one of the 3 pilot sites during the pilot testing phase.
* Pilot site clinicians: nurses, care managers, social workers, and physicians who are employed/provide services in the pilot site.

Exclusion Criteria:

* Patient Exclusion Criteria : Those individuals < 18 years of age, incarcerated, or admitted for reasons other than receipt of intensive care services (e.g. boarders).
* Pilot Site Clinicians Exclusion Criteria: none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of training the staff for the intervention, as measured by percent of staff members completing on-line training | At the completion of the two week training phase which will occur immediately prior to initiating the 3-month pilot of the intervention
  Feasibility of using online training will be assessed by percent of staff members who complete the on-line training during the two week training phase.
Feasibility of patient recruitment at the site, as measured by the volume of eligible patients admitted to the pilot ICU during the pilot phase. | At the conclusion of the 3-month pilot
  Feasibility of recruitment will be assessed by the volume of eligible patient admitted to the pilot ICU.
Adherence to elements of intervention protocol | Throughout the 3 month pilot phase
  Adherence to steps in the intervention protocol for eligible patients will be assessed by review of tracking forms, questions to staff about patient screening and about engagement with family members, and direct observation of staff during interdisciplinary team rounds.
Acceptability of the intervention to clinicians assessed via focus groups | At the conclusion of the 3-month pilot
  Acceptability of the intervention will be evaluated using focus group sessions with physicians, social workers, care managers, and nurses. Using a semi-structured interview guide, we will elicit detailed information about staff satisfaction with the intervention; the clinician experience of participating in the intervention; staff-perceived value of the intervention to patients and families; and suggestions for improvement.
Clinician Satisfaction with the intervention assessed via on-line survey | At the conclusion of the 3-month pilot
  Satisfaction of staff with: 1.) the intervention training and 2.) on-site support, as well as perceived value to patients/families and perceived burden of carrying out the intervention will be evaluated using a multi-item, likert-scale scored online survey sent to physicians, social workers, care managers, and nurses.

SECONDARY OUTCOMES:
Proportion of patients with a family meeting | At the conclusion of the 3-month pilot
  The impact of the intervention will be assessed via the proportion of eligible patients having an interdisciplinary family meeting.
Time elapsed until the first family meeting | At the conclusion of the 3-month pilot
  The impact of the intervention will be assessed via the mean time from enrollment to the first interdisciplinary family meeting.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer B Seaman, PhD,RN,CHPN, Principal Investigator — University of Pittsburgh School of Nursing
Locations (2):
- United States (2):
  - Excela Westmoreland Hospital, Greensburg, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
This study will be conducted at sites within two different health systems, Allegheny Health Network and Excela Health, each with their own Institutional Review Board (IRB). The data use agreements with those respective organizations are pending, and we do not yet know the conditions and specifically, if and under what circumstances data sharing will be permitted.
  Provided data sharing is permitted, and in accordance with those agreements, academic collaborators of the Principal Investigator outside of the University of Pittsburgh may have access to participant data collected during the trial, after de-identification. These outside collaborators will obtain their own IRB approval for their role.
Supporting Information: Study Protocol, SAP
Time Frame: These will be made available beginning 9 months and ending 36 months following article publication.
Access Criteria: We will make this data available to collaborators whose proposed use of the data has been approved by an independent review committee.